CLINICAL TRIAL: NCT06022406
Title: Fecal Microbiota Transplantation to Reduce Immune Activation in ART-treated People Living With HIV With Low CD4/CD8 Ratio: The Gutsy Study
Brief Title: Fecal Microbiota Translantation (FMT) to Reduce Inflammation in PLWH: The Gutsy Pilot Study
Acronym: Gutsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jean-Pierre Routy (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Sponsor-Investigator, Jean-Pierre Routy, Clinical Director of the Chronic Viral Illness Service Division of Hematology and Chronic Viral Illness Service Louis Lowenstein Chair in Hematology & Oncology Professor of Medicine, McGill University, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-9477
Record Dates: First submitted 2023-08-04; First posted 2023-09-01 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: HIV-1-infection
Keywords: HIV; Low CD4/CD8 ratio; Dysbiosis
MeSH Terms: conditions — Dysbiosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, placebo-controlled, interventional study
Who Masked: Participant
Masking Description: Prior to study commencement, a statistician will develop a randomization list and prepare sequentially numbered sealed envelopes containing the randomization group assignment. In this single blind study, participants will not know which arm they have been assigned to.
  After screening, upon validation of eligibility, study staff will open the next sequentially numbered envelope to determine which group the study participant has been assigned to. Randomization after screening will allow sufficient time to prepare capsules and have them shipped to the study site before the first treatment visit (Visit 3-Day 0). The randomization group will be recorded on the randomization electronic case report form (eCRF).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT capsules (Experimental): 10 participants taking FMT. The study product consists of fecal microbiota capsules prepared by Dr. Silverman's team in London, Ontario, Canada. Dr. Silverman has received approval from Health Canada to evaluate FMT in patients with metastatic malignant melanoma or with fatty liver within a clinical trial setting (CTA control nos. 235387and 195078 respectively).
  Approximately 30 to 40 capsules will be prepared from 80-100g of healthy human feces from a single healthy donor and administered as a single dose. Capsules will be prepared by a modified method as described by Kao et al, 201747,48 (see Investigator brochure).
  Interventions: Biological: FMT capsules
- Placebo capsules (Placebo Comparator): 10 participants taking Placebo. Placebo capsules contain microcrystalline cellulose, for equivalence in weight and color that will be encapsulated in gelatin capsules. Each capsule will be filled with approximatively 5.5g of microcrystalline cellulose, and encapsulated in size 0 and size 00 capsules.
  Interventions: Biological: Placebo capsules

INTERVENTIONS:
Biological: FMT capsules — Formulation: 80-100g of healthy donor stool processed, frozen and encapsulated in gelatin capsules (modified Kao et al, 2017).
  Arms: FMT capsules
Biological: Placebo capsules — Formulation: microcrystalline cellulose, for equivalence in weight and color, will be encapsulated in gelatin capsules. Each capsule will be filled with approximatively 5.5g of microcrystalline cellulose, and encapsulated in size 0 and size 00 capsules.
  Arms: Placebo capsules

SUMMARY:
The goal of this randomized, single blind, two-armed pilot study is to assess the efficacy of FMT in reducing gut mucosal and systemic inflammation in ART-treated people living with HIV with low CD4/CD8 ratio. The main questions it aims to answer are: •Is there a change in the gut permeability among participants taking FMT compared to placebo? • Has inflammation been reduced by the use of FMT? Ten participants will be randomized to receive FMT in capsules, and another 10 participants will receive placebo capsules containing microcrystalline cellulose. Capsules will be given twice (30 to 40 capsules at each treatment) at 3 weeks interval, to ensure engraftment. In an optional substudy, participants will be asked to undergo colonoscopy before and 3 months after FMT to assess gut inflammation and HIV reservoir size in colon biopsies. Researchers will compare the FMT arm and the Placebo arm to see if there are differences in gut permeability and inflammation.

DETAILED DESCRIPTION:
Background: HIV infection is characterized by a rapid mucosal CD4 T-cell depletion and early epithelial gut damage. People living with HIV (PLWH) have an abnormal gastrointestinal landscape characterized by villous atrophy, crypt hyperplasia, loosened tight junctions, gastrointestinal inflammation and increased intestinal permeability. Despite long-term antiretroviral therapy (ART), gut mucosa damage remains in PLWH. Increased gut permeability allows the translocation of microbial products into the mucosa and the blood. This process, called microbial translocation, has been associated with increased inflammation and the development of non-AIDS events such as cardiovascular diseases, neurocognitive dysfunction and some cancers in ART-treated PLWH.

Gut damage and persistent inflammation were associated with the modification of the gut microbiota, called dysbiosis, which persists in PLWH under ART. Hence, therapies targeting the gut mucosa are a must.

Minor changes were obtained with Lactobacillus-based probiotics aiming at balancing microbiota composition in PLWH. A promising intervention is the use of fecal microbial transplantation (FMT), which consist of delivering stool microbiota from a donor by upper-endoscopy in the stomach or colonoscopy. More recently, oral delivery of encapsulated stool preparation was shown to lead to a more stable engraftment of the donor's microbiota. FMT was primarily used to eliminate Clostridium difficile infection. FMT is not commonly used in PLWH, but macaque models gave promising results with reduced gut inflammation post FMT in SIV-infected monkeys.

Objectives: To assess, before and after FMT, in the FMT compared to place group:

* Plasma levels of gut damage markers (Intestinal Fatty acid Binding protein) and the new marker of gut permeability Regenerating Islet Derived protein 3 α (REG3α).
* Inflammatory cytokines and T and Myeloid cell activation in blood and colon biopsies
* Changes in stools microbiota composition
* Changes in mucosal and blood HIV reservoir size
* Safety of FMT

Methods: To perform a randomized, single blind, two-armed pilot study in HIV-infected ART treated participant with a low CD4/CD8 ratio which are at higher risk of inflammation and dysbiosis. Ten participants will be randomized to receive FMT in capsules, and another 10 will receive placebo capsules containing microcrystalline cellulose. Capsules will be given twice (30 to 40 capsules at each treatment) at 3 weeks interval, to ensure engraftment. Safety will be assessed. In an optional substudy, participants will be asked to undergo colonoscopy before and 3 months after FMT to assess gut inflammation and HIV reservoir size in colon biopsies.

Anticipated results: We expect that FMT will reduce gut mucosal and systemic inflammation. This study should provide sufficient results for calculation of power in a larger scale trial in PLWH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults ≥18 years of age.
2. Documented HIV-1 infection by Western Blot, Enzyme Immuno Assay (EIA) or viral load assay.
3. On ART for at least 3 years, and stable ART regimen (same prescription) for at least 3 months.
4. Undetectable viral load < 50 copies/ml for the past 3 years. Viral blips below 200 copies/ml, are allowed if preceded and followed by a HIV viremia below 50 copies/ml.
5. CD4 count between greater than 200 cells/µL and a CD4/CD8 ratio below 1 to select people with higher risks of inflammatory non-AIDS comorbidities and dysbiosis.
6. Able to communicate adequately in either French or English.
7. Able and willing to provide written informed consent prior to screening.
8. Women of childbearing potential must have a negative serum pregnancy test at Screening
9. Women of childbearing potential must agree to use one of the following approved methods of birth control while in the study and until 2 weeks after completion of the study (See Section 7.1):

   1. Complete abstinence from penile-vaginal intercourse from the screening period until 2 weeks after study completion.
   2. Double barrier method (acceptable barrier methods include diaphragm, coil, contraceptive foam, sponge with spermicide, or condom).
   3. Oral, injectable or implant contraceptives plus one barrier method.
   4. Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion) plus one barrier method.
   5. Male partner sterilization confirmed prior to the female participant's entry into the study; this male is the sole partner for that participant.
   6. Approved hormonal contraception, started at least 30 days before screening, preferably with one barrier method.
   7. Another method approved by the Investigator with published data showing that the expected failure rate is <1% per year preferably with one barrier method.
10. Women of non-child-bearing potential as defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.
11. Sexually active men with a female partner of childbearing potential must agree to one of the following methods of birth control (See Section 7.1):

    1. The use of at least one barrier method of contraception (e.g. condom) with a female partner using a second approved method of contraception (IUD, hormonal contraceptive pill, diaphragm, spermicide, etc.) during the study and until two weeks after study completion.
    2. Have had a successful vasectomy.
    3. Be confirmed sterile. Any contraception method must be used consistently, in accordance with this study protocol, and for the duration of the study until two weeks after study completion.

Exclusion Criteria:

1. Known allergy/hypersensitivity Polyethylene glycol.
2. Current AIDS-related event or serious health condition including systemic infections in the last 3 months.
3. Severe systemic diseases (e.g. uncontrolled hypertension, chronic renal failure), or active uncontrolled infections.
4. Co-infection with active Hepatitis B or C Virus.
5. Current use or have used in the past 3 months: immune-modulatory agents, prophylactic antibiotics45/antibiotics, or Morphine as these drugs modulate gut microbiota.
6. Diagnosis of diabetes mellitus (HbA1c≥6.5%) as defined by the Canadian Clinical Practice Guidelines for the Prevention and Management of Diabetes46.
7. Recent changes in dietary habits, intermittent fasting, chronic constipation or laxative use as these can affect gut microbiota.
8. Psychiatric or cognitive disturbance or any illness that could preclude compliance with the study.
9. Current participation in an experimental therapy study or receipt of experimental therapy within the last 6 months.
10. Women who are planning to become or who are pregnant, or breast-feeding.
11. A score of higher than 8 on a Full AUDIT questionnaire at the screening visit, suggesting an alcohol abuse problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
REG3α levels | 12 weeks
  Changes in plasma REG3α levels will be measured as markers of gut permeability

SECONDARY OUTCOMES:
Safety of FMT | 12 weeks
  Safety of FMT measured by evaluating adverse events.
Tolerability of FMT | 12 weeks
  tolerability of FMT measured by evaluating adverse events.
Changes in plasma levels of gut damage markers | 12 weeks
  Changes in plasma levels of gut damage markers (I-FABP)
Changes in plasma levels of gut damage markers | 12 weeks
  Changes in plasma levels of gut damage markers (LPS).
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  Changes in Plasma levels of (1-3)-β-D-Glucan will be measured by Multiplex or ELISA.
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-1β will be measured by Multiplex or ELISA.
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-6 will be measured by Multiplex or ELISA.
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-8 will be measured by Multiplex or ELISA.
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  -Changes in Plasma levels of IP-10 will be measured by Multiplex or ELISA.
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-17A and F will be measured by Multiplex or ELISA.
Changes in Plasma levels of pro-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-22 will be measured by Multiplex or ELISA.
Changes in Plasma levels of anti-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-10 will be measured by Multiplex or ELISA.
Changes in Plasma levels of anti-inflammatory markers | 12 weeks
  Changes in Plasma levels of IL-37 will be measured by Multiplex or ELISA.
Changes in T cell activation in blood | 12 weeks
  Changes in T cell activation in blood, as assessed by flow cytometry expression of HLA-DR
Changes in T activation in blood | 12 weeks
  Changes in T cell activation in blood, as assessed by flow cytometry expression of CD38
Changes in myeloid cell activation in blood | 12 weeks
  Changes in myeloid cell activation in blood, as assessed by flow cytometry expression of CD83
Changes in myeloid cell activation in blood | 12 weeks
  Changes in myeloid cell activation in blood, as assessed by flow cytometry expression of CD86

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Berini, Dr., Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Chronic Viral Illness Service, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Isnard S, Berini CA, Parvathy SN, Feng H, Aiyana O, Royston L, Mabanga T, Lakatos PL, Bessissow T, Klein MB, Lebouche B, Costiniuk CT, Routy B, Silverman MS, Routy JP. Fecal microbiota transplantation to reduce immune activation in ART-treated people with HIV with low CD4/CD8 ratio: protocol for the single-blind, randomized, placebo-controlled Gutsy study (CIHR/CTN PT038). Trials. 2025 Dec 13. doi: 10.1186/s13063-025-09345-0. Online ahead of print. PMID 41390455